CLINICAL TRIAL: NCT03840161
Title: Evaluation of the CNOGA TensorTip COMBO GLUCOMETER (CoG) During Standardized Meal Test and Consecutive Home Use by Patients With Diabetes Mellitus
Brief Title: Use of CoG by Patients With Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Sciema UG (Other)
Collaborators: Cnoga Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNG-NGM-003
Record Dates: First submitted 2018-07-21; First posted 2019-02-15 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus Type 1; Diabetes mellitus Type 2; blood glucose self-testing; non-invasive tissue glucose prediction; optical pain-free glucose testing
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: non-invasive tissue glucose prediction — Generation of non-invasive and invasive glucose readings for comparison with a standard laboratory reference glucose determination method (YSI glucose analyzer)
  Other Names: invasive blood glucose measurement

SUMMARY:
The CNOGA Combo Glucometer (CoG) employs an invasive glucose meter using blood glucose teststrips and requiering a capillary blood sample obtained from a fingerstick and in addition, a non-invasive optical component for prediction of tissue glucose at the fingertip. In this study, participants will use both devices during meal tests and also at home during routine care. The results from the device will be compared to a standard reference method and will be used to determine the accuracy of the two device components.

DETAILED DESCRIPTION:
The trial starts with a screening and training visit (V1). This is followed by an individual calibration period for the non-invasive device component by means of multiple parallel measurements with the invasive and the noninvasive device component. This will be done by the participants at home. Thereafter, the participants will come to the study site and will ingest a standardized meal (V2). Blood will be drawn for assessment of HbA1c and biochemical safety parameters. During the next 3 hours, 11 fingersticks will be made to obtain capillary blood samples for comparator readings with the two CoG components and with a laboratory reference method (YSI gucose analyzer). The patients will now continue to use the devices at home for three months, but are not allowed to use any CoG result for treatment decisions. In an interim visit after 6 weeks (V3), blood will be drawrn for HbA1c and biochemical safety parameters and three comparison measurements will be made with the CoG device components and the laboratory reference method. At the final visit after 12 weeks (V4), the procedures of the first meal test visit (V2) will be repeated, which conludes that study. In addition, the participants will be asked to complete a device satisfaction questionnaire at V2, V3, and V4.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or Type 2 diabetes of Afro-American, Hispanic, or Asian-American origin
* Subjects who are able to provide informed consent (by him/herself or by his/her guardian);
* 18 years old and above;
* HbA1c < 10 %
* Anatomically suitable finger as determined by the clinical investigator and detailed in section 4

Exclusion Criteria:

* Does not meet inclusion criteria;
* Subjects requiring dialysis;
* Any conditions that may hamper good visual contact between the finger and sensor, such as raised birthmarks, scars and/or tattoos;
* Pregnancy;
* Nursing mothers;
* Any skin injuries on the measured finger;
* Severe disease conditions (cancer etc.)
* Any condition that may prevent patients from successful participation in the trial (in discretion of the investigator)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes mellitus (type 1 or type 2, any treatment) of other than caucasian origin, who are experienced with performing blood glucose self-testing.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
CoG accuracy in measuring glucose levels (non-invasively) during a standardized meal experiment. | Experiment will be performed twice within 3 months
  Comparison of non-invasive CoG device measurements (tissue glucose in mg/dL) with the results of a standard laboratory reference method (YSI glucose analyzer, blood glucose in mg/dL) by consensus-error grid analysis
CoG accuracy in monitoring glucose levels (invasively) during a standardized meal experiment. | Experiment will be performed twice within 3 months
  Comparison of CoG invasive device readings (blood glucose in mg/dL) with the results of a standard laboratory reference method (YSI glucose analyzer, blood glucose in mg/dL) by consensus-error grid analysis

SECONDARY OUTCOMES:
Impact of the CoG on long-term (three month) glycemic control (HbA1c using standard laboratory procedures) in patients with type 1 and 2 diabetes | 3 months
  Change in HbA1c from baseline after 6 weeks and 12 weeks
Treatment satisfaction questionnaire | 3 months
  Change in device satisfaction questionnaire score after 6 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Demircik, PhD, Study Director — Sciema UG
Locations (1):
- Mills-Penisnsula Medical Center, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No